CLINICAL TRIAL: NCT02760342
Title: ASP015K Pharmacokinetic Study: Evaluation of Drug-Drug Interaction Between ASP015K and Metformin
Brief Title: A Drug Interaction Study to Evaluate the Pharmacokinetics of ASP015K and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 015K-CL-PK20
Record Dates: First submitted 2016-05-01; First posted 2016-05-03 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Metformin; Drug-drug interaction; ASP015K
MeSH Terms: interventions — peficitinib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP015K and Metformin (Experimental): Subjects will receive a single oral dose of metformin on Days 1 and 10, a single dose of ASP015K on Day 3 and multiple doses of ASP015K once daily Day 5 to Day 11. Subjects will receive a single dose of metformin and ASP015K concurrently on Day 10.
  Interventions: Drug: peficitinib; Drug: Metformin

INTERVENTIONS:
Drug: peficitinib — Oral
  Other Names: ASP015K
Drug: Metformin — Oral

SUMMARY:
The objective of this study is to evaluate the pharmacokinetic interactions between ASP015K and metformin in healthy non-elderly male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight at screening: ≥ 50.0 kg, < 80.0 kg
* BMI at screening: ≥ 17.6, < 26.4
* Subjects who agree to use highly effective contraception as consisting of two forms of birth control (at least one of which must be a barrier method) from getting informed consent through 90 days after the final study drug administration.
* Subjects who agree NOT to donate sperm from getting informed consent through 90 days after the final study drug administration.

Exclusion Criteria:

* Subjects who received or are scheduled to receive any investigational drugs in other clinical trials or post-marketing studies within 120 days before screening test or during the screening test to the hospital admission (Day -1).
* Subjects who received or is scheduled to receive any medications (including over-the-counter drugs) within seven days before the hospital admission (Day -1).
* Subjects who received ASP015K or metformin previously.
* Subjects who have a habit of excessive alcohol drinking or smoking.
* Any deviation from the normal range of blood pressure, pulse, body temperature, or 12-lead ECG at screening or on the day of hospital admission (Day -1).
* Subjects who meet any of the following criterion for laboratory tests at screening or on the day of hospital admission (Day -1). Normal ranges of each test specified at the study site or test/assay organization will be used as the normal ranges in this study.
* Subjects with a complication or history of drug allergies.
* Subjects who have a history of clinically serious allergy, which induces generalized urticaria or anaphylactic shock requiring hospital admission.
* Subjects with a complication or history of hepatic disease, renal disease, cardiac disease, congenital short QT syndrome, respiratory disease , gastrointestinal disease.
* Subjects with a history of gastrointestinal resection.
* Subjects who developed upper gastrointestinal symptoms within seven days before the hospital admission (Day -1).
* Subjects with a complication or history of endocrine disease, cerebrovascular disease, malignant tumor, lymphatic disease , lactic acidosis.
* Subjects who apply to any of the concerns with regard to tuberculosis.
* Subjects who apply to any of the concerns with regard to infection other than tuberculosis.
* Subjects with vaccination of live vaccines or live attenuated vaccines within 56 days before the hospital admission (Day -1).

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2016-06-26 (Actual); Study Completion 2016-06-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of metformin in plasma: AUCinf | Up to Day 12
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameter of metformin in plasma: Cmax | Up to Day 12
  Cmax: Maximum concentration
PK parameter of metformin in plasma: AUClast | Up to Day 12
  AUClast: Area under the concentration-time curve from the time of dosing to the last measurable concentration

SECONDARY OUTCOMES:
PK parameter of metformin in plasma: CL/F | Up to Day 12
  CL/F: Apparent total systemic clearance
PK parameter of metformin in plasma: t1/2 | Up to Day 12
  t1/2: Terminal elimination half-life
PK parameter of metformin in plasma: tmax | Up to Day 12
  tmax: Time of Cmax
PK parameter of metformin in plasma: Vz/F | Up to Day 12
  Vz/F: Apparent volume of distribution during the terminal elimination phase
PK parameter of metformin in urine: Aelast | Up to Day 12
  Aelast: Amount of metformin excreted into the urine from the time of dosing to the last measurable concentration
PK parameter of metformin in urine: Aelast% | Up to Day 12
  Aelast%: Percent of metformin excreted into the urine from the time of dosing to the last measurable concentration
PK parameter of metformin in urine: CLR | Up to Day 12
  CLR: Renal clearance
PK parameter of ASP015K in plasma: AUCinf | Up to Day 12
PK parameter of ASP015K in plasma: AUClast | Up to Day 12
PK parameter of ASP015K in plasma: AUCtau | Up to Day 12
  AUCtau: Area under the concentration-time curve from the time of dosing to the start of the next dosing interval
PK parameter of ASP015K in plasma: CL/F | Up to Day 12
PK parameter of ASP015K in plasma: Cmax | Up to Day 12
PK parameter of ASP015K in plasma: Ctrough | Up to Day 12
  Ctrough: Concentration immediately prior to dosing at multiple dosing
PK parameter of ASP015K in plasma: PTR | Up to Day 12
  PTR: Peak trough ratio
PK parameter of ASP015K in plasma: Rac | Up to Day 12
  Rac: accumulation ratio
PK parameter of ASP015K in plasma: t1/2 | Up to Day 12
PK parameter of ASP015K in plasma: tmax | Up to Day 12
PK parameter of ASP015K in plasma: Vz/F | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: AUCinf | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: AUClast | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: AUCtau | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: Cmax | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: Ctrough | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: PTR | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: Rac | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: t1/2 | Up to Day 12
PK parameter of metabolites of ASP015K in plasma: tmax | Up to Day 12
Safety assessed by Adverse events | Up to 17 days after first study drug dosing
Number of participants with abnormal vital signs and/or adverse events related to treatment | Up to 17 days after first study drug dosing
Number of participants with abnormal laboratory values and/or adverse events related to treatment | Up to 17 days after first study drug dosing
Number of participants with abnormal standard 12-lead ECG and/or adverse events related to treatment | Up to 17 days after first study drug dosing
  ECG: Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Kagoshima, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028